# **Cover Page for Statistical Analysis Plan**

| Sponsor name: | Novo Nordisk A/S |
|---|---|
| NCT number | NCT05259033 |
| Sponsor trial ID: | NN1535-4592 |
| Official title of study: | A 52-week study comparing the efficacy and safety of once weekly IcoSema and once weekly semaglutide, both treatment arms with or without oral anti-diabetic drugs, in participants with type 2 diabetes inadequately controlled with a GLP-1 receptor agonist. COMBINE 2 |
| Document date: | 23 June 2022 |

Statistical Analysis Plan Study ID: NN1535-4592


Date: Version: Status: Page: 23 June 2022 5.0 Final


23 June 2022 Novo Nordisk

# Statistical Analysis Plan

A 52-week study comparing the efficacy and safety of once weekly IcoSema and once weekly semaglutide, both treatment arms with or without oral anti-diabetic drugs, in participants with type 2 diabetes inadequately controlled with a GLP-1 receptor agonist. COMBINE 2

Substance: IcoSema (insulin icodec and semaglutide)

23 June 2022 5.0 Final 2 of 27

# **Table of contents**

| | | | | Page |
|---|---|---|---|---|
| | | | S | |
| V | ersion | History | | 4 |
| 1 | Intro | duction. | | 5 |
| | 1.1 | | ves, Endpoints, and Estimands | |
| | | 1.1.1 | Objectives | |
| | | | 1.1.1.1 Primary objective | 5 |
| | | | 1.1.1.2 Secondary objectives | |
| | | 1.1.2 | Endpoints | |
| | | | 1.1.2.1 Primary endpoint | |
| | | | 1.1.2.2 Secondary endpoints | |
| | | | 1.1.2.2.1 Supportive secondary endpoints | |
| | | 1.1.3 | Estimands | |
| | | | 1.1.3.1 Primary Estimand | |
| | 1.0 | C4- 4- F | 1.1.3.2 Supportive Secondary Estimands | |
| | 1.2 | • | Design | |
| 2 | Stati | stical Hy | potheses | 8 |
| | 2.1 | Multipl | icity Adjustment | 8 |
| 3 | Anal | vsis Sets | | 8 |
| | | • | | |
| 4 | Stati<br>4.1 | | alyses | |
| | 4.1 | | Considerations | |
| | 4.2 | 4.2.1 | Definition of Endpoint | |
| | | 4.2.1 | Main Analytical Approach | |
| | | 4.2.3 | Sensitivity Analysis | |
| | | 4.2.4 | Supplementary Analysis | |
| | 4.3 | | ary Estimands Analyses | |
| | | 4.3.1 | Supportive Secondary Estimands | |
| | | | 4.3.1.1 Supportive Secondary Efficacy Estimands | |
| | | | 4.3.1.1.1 Change in body weight from baseline week 0 (V2) to week 52 (V54) | |
| | | | 4.3.1.1.2 Change in fasting plasma glucose (FPG) from baseline week 0 | |
| | | | (V2) to week 52 (V54) | 12 |
| | | | 4.3.1.2 Supportive Secondary Safety Estimands | |
| | | | 4.3.1.2.1 Hypoglycaemic episodes | 12 |
| | 4.4 | Explora | tory Estimands Analysis | 13 |
| | 4.5 | | afety Analysis | |
| | | 4.5.1 | Hypoglycaemic episodes | |
| | | 4.5.2 | Relative change in lipids from baseline week 0 (V2) to week 52 (V54) | |
| | | 4.5.3 | Change in vital signs from baseline week 0 (V2) to week 52 (V54) | |
| | | 4.5.4 | Anti-insulin icodec antibodies | |
| | 1.0 | 4.5.5 | Record selection | |
| | 4.6 | | analyses | |
| | | 4.6.1 | Other Variables and/or Parameters | 15 |
| | | | (V54)(V54) | 15 |
| | | | 4.6.1.2 Achievement of targets | |
| | | 4.6.2 | Pharmacokinetic modelling | |
| | 4.7 | | Analysis | |
| | 4.8 | | s to Protocol-planned Analysis | |

1.0

Statistical Analysis Plan Date: 23 June 2022 Novo Nordisk Study ID: NN1535-4592 Version: 5.0 CONFIDENTIAL Status: Final Page: 3 of 27 4.9 6.2 6.3 

| Statistical Analysis Plan Study ID: NN1535-4592 CONFIDENTIAL | Date:<br>Version:<br>Status:<br>Page: | 23 June 2022 <b>Novo Nordisk</b> 5.0 Final 4 of 27 |
|---|---|---|
|---|---|---|

# **Version History**

This Statistical Analysis Plan (SAP) for study NN1535-4592 is based on the protocol version 7.0 dated 10May2022.

| SAP Version | Date | Change | Rationale |
|---|---|---|---|
| 1.0 | 23Jun2021 | Not Applicable | Original version |
| 2.0 | 02Jul2021 | Reference to protocol version updated | The protocol was updated to version 2.0. |
| 3.0 | 10Aug2021 | Reference to protocol version updated | The protocol was updated to version 4.0. |
| 4.0 | 16Mar2022 | Clarification of analysis | The offset in a statistical analysis has been clarified. |
| 5.0 | 23Jun2022 | Reference to protocol<br>version updated<br>Addition of Hungary and<br>removal of Ukraine in the<br>definition of regions | To reflect the new country allocation for the study |

23 June 2022 5.0 Final


23 June 2022 | Novo Nordisk

## 1 Introduction

This SAP is based on the protocol: A 52-week study comparing the efficacy and safety of once weekly IcoSema and once weekly semaglutide, both treatment arms with or without oral anti-diabetic drugs, in participants with type 2 diabetes inadequately controlled with a GLP-1 receptor agonist. COMBINE 2. This SAP include details on analysis of secondary estimands related to supportive secondary endpoints. There are no changes to the analyses described in the protocol, however additional information has been included in case of insufficient data for meaningful imputation of missing data for the primary analysis. The SAP also contains specification of additional derivations and analyses.

#### 1.1 Objectives, Endpoints, and Estimands

## 1.1.1 Objectives

#### 1.1.1.1 Primary objective

To confirm superiority of once weekly IcoSema compared with once weekly semaglutide, both treatment arms with or without OADs, in terms of glycaemic control measured by change in HbA<sub>1c</sub> from baseline after 52 weeks in participants with T2D inadequately controlled a GLP-1 receptor agonist.

#### 1.1.1.2 Secondary objectives

To compare parameters of glycaemic control and safety of once weekly IcoSema with once weekly semaglutide, both treatment arms with or without OADs, in participants with T2D inadequately controlled with a GLP-1 receptor agonist.

#### 1.1.2 Endpoints

#### 1.1.2.1 Primary endpoint

| Endpoint title | Time frame | Unit |
|---|---|---|
| Change in HbA <sub>1c</sub> | From baseline week 0 (V2) to week 52 (V54) | %-point |

#### 1.1.2.2 Secondary endpoints

## 1.1.2.2.1 Supportive secondary endpoints

#### Secondary efficacy endpoints

| <b>Endpoint title</b> | Time frame | Unit |
|---|---|---|
| Change in fasting plasma glucose (FPG) | From baseline week 0 (V2) to week 52 (V54) | mmol/L |
| Change in body weight | From baseline week 0 (V2) to week 52 (V54) | Kg |

Status: Page:

5.0 Final 6 of 27

#### Secondary safety endpoints

| Endpoint title | Time frame | Unit |
|---|---|---|
| Number of clinically significant<br>hypoglycaemic episodes (level 2)<br>(<3.0 mmol/L (54 mg/dL), confirmed by<br>BG meter) or severe hypoglycaemic<br>episodes (level 3) | From baseline week 0 (V2) to week 57 (V56) | Number of episodes |
| Number of clinically significant hypoglycaemic episodes (level 2) (<3.0 mmol/L (54 mg/dL), confirmed by BG meter) | From baseline week 0 (V2) to week 57 (V56) | Number of episodes |
| Number of severe hypoglycaemic episodes (level 3) | From baseline week 0 (V2) to week 57 (V56) | Number of episodes |

#### 1.1.3 Estimands

#### 1.1.3.1 **Primary Estimand**

The primary estimand is described by the following 5 attributes:

- Treatment condition: The effect of randomised treatment (titration of once weekly IcoSema versus fixed dose escalation of once weekly semaglutide 1 mg) with or without OAD(s), regardless of initiation of non-randomised insulin treatment or additional antidiabetic treatments for more than 2 weeks and adherence to randomised treatment
- Population: T2D inadequately controlled with a GLP-1 receptor agonist
- Endpoint: Change in HbA<sub>1c</sub> from baseline to week 52
- Remaining ICEs: None. The two intercurrent events are captured under treatment condition and handled as follows:
  - o Initiation of non-randomised insulin treatment or additional antidiabetic treatments for more than 2 weeks by the treatment policy strategy
  - Discontinuation of randomised treatment for any reason by the treatment policy strategy
- Population-level summary: Difference in mean changes from baseline

#### 1.1.3.2 **Supportive Secondary Estimands**

#### Estimand related to change in body weight from baseline to week 52

The estimand is the same as for the primary estimand except with the endpoint attribute specified as: Change in body weight from baseline to week 52.

#### Estimand related to change in fasting plasma glucose (FPG) from baseline to week 52

The estimand is described by the following 5 attributes:

Treatment condition: The effect of randomised treatment (titration of once weekly IcoSema versus fixed dose escalation of once weekly semaglutide 1 mg) with or without OAD(s),


23 June 2022 | Novo Nordisk

regardless of initiation of non-randomised insulin treatment or additional antidiabetic treatments for more than 2 weeks and had all participants adhered to randomised treatment

- Population: T2D inadequately controlled with a GLP-1 receptor agonist
- Endpoint: Change in fasting plasma glucose (FPG) from baseline to week 52
- Remaining ICEs: None. The two intercurrent events are captured under treatment condition and handled as follows:
  - o Initiation of non-randomised insulin treatment or additional antidiabetic treatments for more than 2 weeks by the treatment policy strategy
  - o Discontinuation of randomised treatment for any reason by the hypothetical strategy
- Population-level summary: Difference in mean

#### Estimands related to supportive secondary safety endpoints

Supportive secondary estimands related to supportive secondary safety endpoints are similar to the estimand specified for FPG except for the endpoints attributes being specified as the respective supportive secondary safety endpoint and the population-level summary attributed being specified as "Rate ratio".

#### 1.2 Study Design

This is an interventional, multi-national, multi-centre, randomised, 52-week, open label, parallel group, treat-to-target/dose escalation, confirmatory study with two treatment arms. The study investigates the efficacy and safety of treatment with once weekly IcoSema compared to once weekly semaglutide, both treatment arms with or without OADs, in participants with T2D inadequately controlled with a GLP-1 receptor agonist.

The study duration is approximately 59 weeks and consists of:

- an up to 2 weeks screening period
- a 52-week treatment period
- a 5-week follow-up period

The overall study design is outlined in <u>Figure 1-1</u>. For further details see the study protocol.

Figure 1-1 Study design



| Statistical Analysis Plan<br>Study ID: NN1535-4592 | CONFIDENTIAL | Date:<br>Version:<br>Status:<br>Page: | 23 June 2022 <b>N</b><br>5.0<br>Final<br>8 of 27 | lovo Nordisk |
|---|---|---|---|---|
|---|---|---|---|---|

# 2 Statistical Hypotheses

The primary objective is to show that IcoSema is superior to semaglutide in terms of change in HbA<sub>1c</sub> (%) from baseline week 0 (V2) to week 52 (V54).

Formally, let D be the mean treatment difference 'IcoSema' minus 'semaglutide' of the change in  $HbA_{1c}$  (%) from baseline week 0 (V2) to week 52 (V54). The null-hypothesis of IcoSema not being superior will be tested against the alternative hypothesis of superiority as given by

$$H_0$$
:  $D \ge 0\%$  against  $H_A$ :  $D < 0\%$ 

Superiority will be considered confirmed if the upper bound of the two-sided 95% confidence interval for D is strictly below 0 %.

#### 2.1 Multiplicity Adjustment

Not applicable for this study.

## 3 Analysis Sets

The following populations are defined:

| Participant analysis set | Description |
|---|---|
| Full analysis set | All randomised participants. Participants will be included in the analyses |
| | according to the planned randomised treatment. |
| Safety analysis set | All randomised participants who are exposed to randomised treatment. |
| | Participants will be included in the analyses according to the randomised |
| | treatment they actually received. |

The following data points sets are defined:

| Data points sets | Description |
|---|---|
| In-study | All data from randomisation until the last date of any of the following: |
| | The last direct participant-site contact |
| | Withdrawal for participants who withdraw their informed consent |
| | The last participant-investigator contact as defined by the investigator |
| | for participants who are lost to follow-up (i.e. possibly an unscheduled |
| | phone visit) |
| | <ul> <li>Death for participants who die before any of the above</li> </ul> |
| On-treatment | All data from the date of first dose of randomised treatment as recorded on the |
| | eCRF until the first date of any of the following: |
| | • The last follow-up visit (V56) |
| | • The last date on randomised treatment +6 weeks (corresponding to 5 |
| | weeks after the end of the dosing interval for both treatment arms) |
| | The end-date for the in-study data points sets |

The on-treatment data points set represent data collected in the period in which a participant is considered exposed to randomised treatment.

Baseline assessments are always included in the in-study and on-treatment data points sets.

| Statistical Analysis Plan<br>Study ID: NN1535-4592 | CONFIDENTIAL | Date:<br>Version:<br>Status: | 23 June 2022<br>5.0<br>Final | Novo Nordisk |
|---|---|---|---|---|
| | | Page: | 9 of 27 | |

The full analysis set and the in-study data points set will be used to estimate the primary estimand.

Efficacy will be evaluated using the full analysis set and in-study data points set. Whereas safety will be evaluated using the on-treatment data points set with descriptive statistics being based on the safety analysis set and statistical analyses being based on full analysis set unless otherwise specified.

## 4 Statistical Analyses

#### 4.1 General Considerations

Baseline is defined as information collected at week 0 (V2). In case a measurement is not available at week 0 (V2) the most recent measurement prior to week 0 (V2) will be used as baseline.

Presentation of results from a statistical analysis will include the estimated mean treatment difference (or ratio) presented together with the two-sided 95% confidence interval and the corresponding two-sided p-value.

In the statistical models, explanatory factors will be coded as follows:

- Randomised treatment: Once weekly IcoSema, Once weekly semaglutide
- Region: Asia, Europe, North America, Other

The regions will be defined as follows:

- Asia: Japan, China, Taiwan
- Europe: France, Greece, Slovakia, Switzerland, Sweden, Hungary
- North America: United States, Canada
- Other: Russia, Israel, Brazil

#### 4.2 Primary Estimand Analysis

#### 4.2.1 Definition of Endpoint

The primary endpoint is change in HbA<sub>1c</sub> from baseline week 0 (V2) to week 52 (V54).

## 4.2.2 Main Analytical Approach

The primary endpoint is change in HbA<sub>1c</sub> from baseline week 0 (V2) to week 52 (V54).

The estimand (see Section 1.1.3.1), will be estimated based on the full analysis set using the instudy data points set which includes all  $HbA_{1c}$  measurements obtained at week 52 (V54) especially measurements from participants experiencing intercurrent events. The imputation approach for the primary estimand is a multiple imputation similar to the one described by McEvoy.

 Missing HbA<sub>1c</sub> measurements at week 52 (V54) for participants experiencing intercurrent events will be imputed from participants experiencing intercurrent events and have a measurement at week 52 (V54) in each treatment arm.

• Missing HbA<sub>1c</sub> measurements at week 52 (V54) for participants not experiencing intercurrent events are imputed from available measurements at week 52 (V54) from participants not experiencing intercurrent events in each treatment arm.

The multiple imputation approach will be done the following way:

- Imputation: An ANCOVA model for change in HbA<sub>1c</sub> from baseline week 0 (V2) to week 52 (V54) for participants experiencing intercurrent events and have a measurement at week 52 (V54) with randomised treatment as fixed factor, last available planned on-treatment HbA<sub>1c</sub> observation without initiation of non-randomised insulin treatment or additional anti-diabetic treatments for more than 2 weeks, the time point (study day) of last available planned ontreatment HbA<sub>1c</sub> observation without initiation of non-randomised insulin treatment or additional anti-diabetic treatments for more than 2 weeks and baseline HbA<sub>1c</sub> as covariate. If participants not experiencing intercurrent events are missing measurements at week 52 (V54) an ANCOVA model will be defined in a similar way using available data from participants not experiencing intercurrent events. The estimated parameters, and their variances, from the imputation models will be used to impute missing HbA<sub>1c</sub> measurements at week 52 (V54). This will be done 1000 times and results in 1000 complete datasets.
- For each of the complete data sets, the primary endpoint will be analysed using an ANCOVA model with region and randomised treatment as fixed factors, and baseline HbA<sub>1c</sub> as covariate. The estimates and standard deviations for the 1000 data sets will be pooled to one estimate and associated standard deviation using Rubin's rule.<sup>2</sup>
- From the pooled estimate and standard deviation the 95% confidence interval for the treatment difference will be calculated. The corresponding two-sided p-value will also be calculated.

This analysis has the underlying assumption that participants with missing data behave similarly as comparable participants within the same treatment arm i.e. that participants experiencing intercurrent events with missing data at week 52 (V54) behave like participants experiencing intercurrent events with data at week 52 (V54) within the same treatment arm and similar for participants not experiencing intercurrent events.

In case the amount of data for the described imputation model is insufficient for meaningful imputation, the first alternative will be the following:

1. Simplifying the imputation model by removing the following covariates from the imputation model: Last available planned on-treatment HbA<sub>1c</sub> observation without initiation of non-randomised insulin treatment or additional anti-diabetic treatments for more than 2 weeks and the time point (study day) of last available planned on-treatment HbA<sub>1c</sub> observation without initiation of non-randomised insulin treatment or additional anti-diabetic treatments for more than 2 weeks.

If the amount of data for this reduced model is still insufficient for meaningful imputation, the following imputation strategy will be applied instead:

2. Missing values at week 52 (V54) will be imputed with baseline value adding a random error term. This imputation method also includes measurements collected after intercurrent events but is otherwise similar to the imputation method for endpoints where there is no data collection

after discontinuation of randomised treatment as described for change in FPG (see section 4.3.1.1.2).

5.0 Final


Missing HbA<sub>1c</sub> at week 52 (V54) will be summarised by participant randomised treatment completion status.

#### 4.2.3 **Sensitivity Analysis**

The following sensitivity analysis will evaluate the robustness of the results towards the missing data assumption.

For the primary endpoint, a two-dimensional tipping point analysis will be performed where participants having imputed HbA<sub>1c</sub> measurement at week 52 (V54) are assumed to have a worse outcome in the IcoSema arm and a better outcome in the semaglutide arm compared to what was imputed in the primary analysis. This is done by adding or subtracting values  $\Delta_i$  to the imputed HbA<sub>1c</sub> values before analysing the data. The value of  $\Delta_i$  will be varied independently in the two treatment arms. The plausibility of the values of  $\Delta_i$  where the conclusion of the primary analysis change will be evaluated to assess the robustness of the primary analysis results.

#### 4.2.4 **Supplementary Analysis**

The following supplementary analysis addressing a attributable estimand similar to the one described by Darken<sup>3</sup> will be prepared. This estimand aims at estimating the effect of randomised treatment had all participants stayed on the randomised treatment for the entire 52 weeks treatment period. Intercurrent events that are considered adversely related to randomised treatment are considered attributable and are handled with a composite estimand strategy and a hypothetical estimand strategy is used for the remainder intercurrent events and data missing e.g. due to participants being lost to follow-up.

The supplementary analysis will be done the following way:

- Participants experiencing intercurrent events that are considered attributable are identified, see Appendix 3 (section 6.36.3) for split into attributable and none attributable intercurrent events.
- Outcome after intercurrent events which are deemed attributable to randomised treatment are assigned the same unfavourable value in the following way:
  - A mixed-effect model for repeated measurements (MMRM) for change from baseline in HbA<sub>1c</sub> is fitted to data obtained before experiencing intercurrent events. The model include treatment, visit and interaction between treatment and visit as fixed effects, and subject as random effect.
  - The unfavourable value is assigned as the estimated change from baseline from the comparator arm at week 52 (V54) plus the standard deviation of the random intercept multiplied by the 90<sup>th</sup> percentile of the standard normal distribution.
- The remaining missing data is imputed using a similar approach as for the primary analysis.

23 June 2022 5.0 Final 12 of 27

23 June 2022 | Novo Nordisk

#### 4.3 Secondary Estimands Analyses

#### 4.3.1 Supportive Secondary Estimands

#### 4.3.1.1 Supportive Secondary Efficacy Estimands

The following subsections describe how the supportive secondary estimands related to supportive secondary efficacy endpoints (see section 1.1.3.2) will be estimated. The subsections refer to the corresponding supportive secondary endpoint. For calculation of endpoints please see appendix 2, section 6.2.

#### 4.3.1.1.1 Change in body weight from baseline week 0 (V2) to week 52 (V54)

The supportive secondary estimand regarding change in body weight from baseline week 0 (V2) to week 52 (V54) will be estimated using a model similar to the primary analysis above substituting body weight for  $HbA_{1c}$ .

# 4.3.1.1.2 Change in fasting plasma glucose (FPG) from baseline week 0 (V2) to week 52 (V54)

The supportive secondary estimand regarding change in FPG from baseline week 0 (V2) to week 52 (V54) will be estimated using a multiple imputation model as described below.

Missing FPG values at week 52 (V54) (regardless of treatment completion status) for both treatment arms will be imputed with baseline value adding a random error term. The random error term is normally distributed with a standard deviation set equal to the estimated residual standard deviation of an ANCOVA analysis on the last available observation before experiencing intercurrent events. Specifically, the imputations and analyses will be carried out as follows:

- First, an ANCOVA model with region and randomised treatment as fixed factors, and a baseline
  value as a covariate will be fitted to the last available observation before experiencing
  intercurrent events.
- Second, the estimated residual standard deviation, *s*, from this model will be used to impute missing values by the baseline value, adding a random normally distributed term with mean zero and standard deviation *s*. This will be done 1000 times.
- For each of the complete data sets, the endpoint will be analysed using an ANCOVA model with region and randomised treatment as fixed factors, and a baseline value as a covariate. The estimates and SDs for the 1000 data sets will be pooled to one estimate and associated SD using Rubin's rule.<sup>4</sup>
- From the pooled estimate and standard deviation the 95% confidence interval for the treatment difference will be calculated. The corresponding two-sided p-value will also be calculated.

#### 4.3.1.2 Supportive Secondary Safety Estimands

#### 4.3.1.2.1 Hypoglycaemic episodes

The supportive secondary estimands regarding the following supportive secondary safety endpoints will be analysed separately using the method described below:

- Number of clinically significant hypoglycaemic episodes (level 2) (<3.0 mmol/L [54 mg/dL], confirmed by BG meter) or severe hypoglycaemic episodes (level 3) from baseline week 0 (V2) to week 57 (V56)
- Number of clinically significant hypoglycaemic episodes (level 2) (<3.0 mmol/L [54 mg/dL], confirmed by BG meter) from baseline week 0 (V2) to week 57 (V56)
- Number of severe hypoglycaemic episodes (level 3) from baseline week 0 (V2) to week 57 (V56)

For participants who discontinued randomised treatment, the number of episodes in the period where hypoglycaemic episodes are not collected (the period from time of follow-up 2 visit (V56) to planned end of the on-treatment data point set) will be imputed using a multiple imputation technique, assuming that the episode rate pre-follow-up 2 (V56) follows the respective treatment arms rate whilst post-follow-up 2 (V56) episode rate is the rate of the comparator arm. The imputation will be done as follows:

- First, a Bayes negative binomial model with log-link function is fitted to the number of episodes data for participants in the comparator arm to obtain the posterior distribution of model parameters. The model will include region as fixed factor and the logarithm of the time period in which a participant is considered exposed to randomised treatment as offset.
- Second, based on the estimated parameters for the comparator arm in this model, the number of episodes in the missing period will be imputed for participants having discontinued randomised treatment. One thousand (1000) complete dataset are generated by sampling from the estimated distribution.
- For each of the complete datasets, the number of episodes will be analysed using a negative binomial model with log-link function, treatment and region fixed factors and offset as described in step 1 plus the missing period for which the number of episodes have been imputed. The estimates and standard errors for the 1000 data sets will be pooled to one estimate and associated standard deviation using Rubin's rule.<sup>4</sup>
- From the pooled estimate and standard deviation the 95% confidence interval will be calculated and back-transformed to the original scale resulting in a treatment ratio and a 95% confidence interval for the treatment ratio. The corresponding two-sided p-value will also be calculated.

The endpoints are defined as described in Protocol Appendix 7.

#### 4.4 Exploratory Estimands Analysis

Not applicable for this study.

#### 4.5 Other Safety Analysis

The standard safety assessments (AEs, safety laboratory parameters, vital signs, etc.) will be reported descriptively; including any notable changes of clinical interest in laboratory parameters.

23 June 2022 5.0 Final 14 of 27

23 June 2022 | Novo Nordisk

## 4.5.1 Hypoglycaemic episodes

Number of nocturnal clinically significant hypoglycaemic episodes (level 2) (<3.0 mmol/L (54 mg/dL), confirmed by BG meter) or nocturnal severe hypoglycaemic episodes (level 3) from baseline week 0 (V2) to week 57 (V56) will be derived and analysed using the same model as specified for the supportive secondary estimands related to the supportive secondary safety endpoints.

The following derivations will be analysed separately using the model as specified for the supportive secondary estimand related to number of hypoglycaemic episodes substituting the ontreatment data point set with data points from baseline week 0 (V2) to week 52 (V54), and substituting 'follow-up 2 visit (V56)' with 'discontinuation of randomised treatment':

- Number of clinically significant hypoglycaemic episodes (level 2) (<3.0 mmol/L (54 mg/dL), confirmed by BG meter) or severe hypoglycaemic episodes (level 3) from baseline week 0 (V2) to week 52 (V54)
- Number of clinically significant hypoglycaemic episodes (level 2) (<3.0 mmol/L (54 mg/dL), confirmed by BG meter) from baseline week 0 (V2) to week 52 (V54)
- Number of severe hypoglycaemic episodes (level 3) from baseline week 0 (V2) to week 52 (V54)

The derivations is defined as described in Protocol Appendix 7.

## 4.5.2 Relative change in lipids from baseline week 0 (V2) to week 52 (V54)

Relative change in lipids from baseline week 0 (V2) to week 52 (V54) will be analysed separately for each of the lipid parameters (see Protocol Appendix 2) using a model similar to the analysis for change in FPG substituting the respective lipid parameter for FPG. A multiplicative model will be used, i.e. the parameter together with the corresponding baseline value will be log-transformed before analysis. The treatment difference and the 95% confidence interval will be back-transformed to the original scale resulting in a treatment ratio and a 95% confidence interval for the treatment ratio.

#### 4.5.3 Change in vital signs from baseline week 0 (V2) to week 52 (V54)

Change in vital signs (pulse rate, systolic and diastolic blood pressure) from baseline week 0 (V2) to week 52 (V54) will be analysed separately for each of the parameters using a model similar to the analysis for change in FPG substituting the respective vital signs parameter for FPG.

#### 4.5.4 Anti-insulin icodec antibodies

Antibodies will be evaluated using the in-study data points set. The following will be summarised by visit for participants randomised to IcoSema:

- Anti-insulin icodec binding antibodies (positive/negative)
- Anti-insulin icodec antibodies cross-reactivity to human insulin status (positive/negative)
- Anti-insulin icodec antibody titres and change from baseline in anti-insulin icodec antibody titres

The correlation between anti-insulin icodec antibodies titres and actual weekly basal insulin dose, HbA<sub>1c</sub>, and change from baseline in HbA<sub>1c</sub>, respectively, will be illustrated using mean plots by treatment week for quartiles of peak post baseline to week 52 (V54) titre values.

The Spearman's rank correlation coefficient between change in anti-insulin icodec antibodies titres at week 52 (V54) and each of the following assessments will be derived with the corresponding p-value for test of no correlation:

- actual weekly basal insulin dose from week 50 (V52) to week 52 (V54)
- HbA<sub>1c</sub> at week 52 (V54)
- change from baseline in HbA<sub>1c</sub> at week 52 (V54)
- level 2 and level 3 combined hypoglycaemic episodes for episodes in the on-treatment data points set

Number and percentage of participants with "treatment-induced" and "treatment-boosted" anti-insulin icodec antibodies will also be summarised. "Treatment-induced" anti-insulin icodec antibodies are defined as cases in which participants switch from negative anti-insulin icodec antibodies at baseline to positive anti-insulin icodec antibodies during the study. "Treatment-boosted" anti-insulin icodec antibodies are defined as cases in which participants, who have positive anti-insulin icodec antibodies at baseline, experience that anti-insulin icodec antibodies titres increase by at least two 2-fold dilution steps during the study.

#### 4.5.5 Record selection

A re-test at any visit is defined as repeating the same laboratory assessment using new sample material. A re-test may be taken if a participant shows up in a non-fasting state for a laboratory assessment that is to be taken in a fasting condition or when sample material is lost or damaged.

In case of multiple eligible assessments at same planned time point (where only one was planned) only the first value will be selected.

#### 4.6 Other Analyses

#### 4.6.1 Other Variables and/or Parameters

For calculation of derivations please see appendix 2, section 6.2.

#### 4.6.1.1 Change in waist circumference from baseline week 0 (V2) to week 52 (V54)

Change in waist circumference from baseline week 0 (V2) to week 52 (V54) will be analysed using a model similar to the analysis for change in FPG substituting waist circumference for FPG.

#### 4.6.1.2 Achievement of targets

The following derivations will be analysed separately using the method described below:

- Achievement of HbA<sub>1c</sub><7.0% at week 52 (V54) (yes/no)
- Achievement of HbA<sub>1c</sub><7.0% at week 52 (V54) without severe (level 3) or clinically significant hypoglycaemic episodes (level 2) (<3.0 mmol/L (54 mg/dL), confirmed by BG meter) during the prior 12 weeks (yes/no)

- Achievement of HbA<sub>1c</sub><7.0% at week 52 (V54) without severe hypoglycaemic episodes (level 3) during the prior 12 weeks (yes/no)
- Achievement of HbA<sub>1c</sub>≤6.5% at week 52 (V54) (yes/no)
- Achievement of HbA<sub>1c</sub>≤6.5% at week 52 (V54) without severe (level 3) or clinically significant hypoglycaemic episodes (level 2) (<3.0 mmol/L (54 mg/dL), confirmed by BG meter) during the prior 12 weeks (yes/no)
- Achievement of HbA<sub>1c</sub>≤6.5% at week 52 (V54) without severe hypoglycaemic episodes (level
   3) during the prior 12 weeks (yes/no)
- Achievement of HbA<sub>1c</sub><7.0% at week 52 (V54) without body weight gain (yes/no)
- Achievement of HbA<sub>1c</sub><7.0% at week 52 (V54) without body weight gain and severe (level 3) or clinically significant hypoglycaemic episodes (level 2) (<3.0 mmol/L (54 mg/dL), confirmed by BG meter) during the prior 12 weeks (yes/no)
- Achievement of HbA<sub>1c</sub><7.0% at week 52 (V54) without body weight gain and severe hypoglycaemic episodes (level 3) during the prior 12 weeks (yes/no)
- Achievement of HbA<sub>1c</sub>≤6.5% at week 52 (V54) without body weight gain (yes/no)
- Achievement of HbA<sub>1c</sub>≤6.5% at week 52 (V54) without body weight gain and severe (level 3) or clinically significant hypoglycaemic episodes (level 2) (<3.0 mmol/L (54 mg/dL), confirmed by BG meter) during the prior 12 weeks (yes/no)</li>
- Achievement of HbA<sub>1c</sub>≤6.5% at week 52 (V54) without body weight gain and severe hypoglycaemic episodes (level 3) during the prior 12 weeks (yes/no)

See Appendix 2, section 6.2, for further details.

Missing change in  $HbA_{1c}$  at week 52 (V54) and missing change in body weight at week 52 (V54) will be imputed in the same way as for the primary analysis (step 1 in section 4.2.2), substituting body weight for  $HbA_{1c}$  when imputing missing body weight assessments, before deriving the dichotomous outcome. Participants who discontinue randomised treatment will have the dichotomous outcome also evaluating hypoglycaemia set to 'no'. For each of the 1000 complete data sets, the derivation will be analysed using a logistic regression model with region and randomised treatment as fixed factors, and baseline  $HbA_{1c}$  value as a covariate. The estimates and standard deviations for the 1000 data sets will be pooled to one estimate and associated standard deviation using Rubin's rule.<sup>4</sup>

#### 4.6.1.3 Self-measured plasma glucose (SMPG)

Mean pre-breakfast SMPG used for dose adjustment in the IcoSema arm and mean pre-breakfast SMPG in the semaglutide arm will be summarised by visit and randomised treatment. Furthermore, number and percentage of participants achieving mean pre-breakfast SMPG used for dose adjustment in the IcoSema arm and mean pre-breakfast SMPG in the semaglutide arm within range (4.4–7.2 mmol/l) will be presented by visit and randomised treatment.

#### 4.6.1.4 Antidiabetic background medication

Participants experiencing changes to antidiabetic background medication during the study lasting more than 2 weeks will be summarised descriptively by randomised treatment including number and proportion of participants.

23 June 2022 Novo Nordisk 5.0 Final 17 of 27

#### 4.6.2 Pharmacokinetic modelling

Insulin icodec serum concentration data and semaglutide plasma concentration data will be used for population PK analysis. The objective of the population PK analysis is to evaluate the effects of relevant covariates on insulin icodec and semaglutide exposure.

The population PK analysis will be performed by Quantitative Clinical Pharmacology, Novo Nordisk. A more technical and detailed elaboration of the population PK analysis will be given in a modelling analysis plan, which will be prepared before database lock. In brief, previously developed PK models for insulin icodec and semaglutide will be applied. The absorption rate constants in the models will be fixed, and the apparent clearance and volume of distribution parameters will be re-estimated. The covariates of interest will be incorporated into the PK models using criteria which will be specified in the modelling analysis plan.

The population PK analysis will be reported in a separate modelling report, which will not be part of the clinical study report. The individual insulin icodec serum concentration data and the individual semaglutide plasma concentration data will be tabulated in the bioanalytical report.

#### 4.7 **Interim Analysis**

Not applicable for this study.

#### 4.8 **Changes to Protocol-planned Analysis**

There are no changes to the protocol-planned analysis.

#### 4.9 Partial database lock

A partial database lock may be performed at the end of the treatment period for all participants, i.e. after the date of the last participant last treatment visit. The database will be updated after the partial database lock to include remaining safety information. The full database lock will be performed after the date of the last participant last visit.

The analysis of the primary endpoint and all other efficacy endpoints will be performed based on the data from the partial database lock. Analysis of safety data will be performed after the full database lock. This approach is implemented to allow earlier availability of IcoSema to a T2D patient population in need of treatment intensification expected to benefit from an insulin and GLP-1 combination product. A detailed plan for data handling and operational aspects of the partial database lock and the database update will be finalised before the partial database lock.

Statistical Analysis Plan
Study ID: NN1535-4592


Date: 23 June 2022 Version: 5.0
Status: Final Page: 18 of 27

# 5 Sample size determination

Please see the protocol section 9.5.

June 2022 5.0 Final


23 June 2022 Novo Nordisk

# **6 Supporting Documentation**

Statistical Analysis Plan

Study ID: NN1535-4592

## 6.1 Appendix 1: List of abbreviations

| AE | Adverse event |
|--------|----------------------------------------------|
| ANCOVA | Analysis of covariance |
| BG | Blood glucose |
| CGM | Continuous glucose monitoring |
| FPG | Fasting plasma glucose |
| ICE | Intercurrent event |
| MMRM | Mixed-effect model for repeated measurements |
| OAD | Oral anti-diabetic drug |
| PK | Pharmacokinetic |
| SAP | Statistical analysis plan |
| SMPG | Self-measured plasma glucose |
| T2D | Type 2 diabetes mellitus |

## 6.2 Appendix 2: Definition and calculation of endpoints, assessments and derivations

| Type | Title | Time frame | Unit | Details |
|---|---|---|---|---|
| Primary endpoint | Change in HbA <sub>1c</sub> | From baseline<br>week 0 (V2) to<br>week 52 | %-point | The HbA <sub>1c</sub> value at baseline week 0 subtracted from the HbA <sub>1c</sub> value at week 52. |
| Supportive<br>secondary efficacy<br>endpoint | Change in body weight | From baseline<br>week 0 (V2) to<br>week 52 (V54) | Kg | The body weight value at baseline week 0 subtracted from the body weight value at week 52. |
| Supportive secondary efficacy endpoint | Change in fasting plasma glucose (FPG) | From baseline<br>week 0 (V2) to<br>week 52 (V54) | mmol/L | The FPG value at baseline week 0 subtracted from the FPG value at week 52. |
| Supportive secondary safety endpoint | Number of clinically significant hypoglycaemic episodes (level 2) (<3.0 mmol/L (54 mg/dL), confirmed by BG meter) or severe hypoglycaemic episodes (level 3) | From baseline<br>week 0 (V2) to<br>week 57 (V56) | Number of episodes | The count of all clinically significant hypoglycaemic episodes (level 2) (<3.0 mmol/L (54 mg/dL), confirmed by BG meter) or severe hypoglycaemic episodes (level 3) within the time frame. |
| Supportive<br>secondary safety<br>endpoint | Number of clinically significant hypoglycaemic episodes (level 2) (<3.0 mmol/L (54 mg/dL), confirmed by BG meter) | From baseline<br>week 0 (V2) to<br>week 57 (V56) | Number of episodes | The count of all clinically significant hypoglycaemic episodes (level 2) (<3.0 mmol/L (54 mg/dL) confirmed by BG meter) within the time frame. |
| Supportive secondary safety endpoint | Number of severe<br>hypoglycaemic episodes<br>(level 3) | From baseline<br>week 0 (V2) to<br>week 57 (V56) | Number of episodes | The count of all severe hypoglycaemic episodes (level 3) within the time frame. |

| Study ID: NN1535 | -4592 | C | ONFIDENTIAL | Version:<br>Status:<br>Page: | 5.0<br>Final<br>20 of 27 |
|---|---|---|---|---|---|
| Derivation | Number of clin significant hypoglycaemic (level 2) (<3.0 (54 mg/dL), corby BG meter) of hypoglycaemic (level 3) | episodes<br>mmol/L<br>nfirmed<br>or severe | From baseline<br>week 0 (V2) to<br>week 52 (V54) | umber of isodes | The count of all clinically significant hypoglycaemic episodes (level 2) (<3.0 mmol/L (54 mg/dL), confirmed by BG meter) or severe hypoglycaemic episodes (level 3) within the time frame. |
| Derivation | Number of clin<br>significant<br>hypoglycaemic<br>(level 2) (<3.0<br>(54 mg/dL), co<br>by BG meter) | episodes<br>mmol/L | From baseline<br>week 0 (V2) to<br>week 52 (V54) | umber of isodes | The count of all clinically significant hypoglycaemic episodes (level 2) (<3.0 mmol/L (54 mg/dL) confirmed by BG meter) within the time frame. |
| Derivation | Number of seven hypoglycaemic (level 3) | | From baseline<br>week 0 (V2) to<br>week 52 (V54) | imber of isodes | The count of all severe hypoglycaemic episodes (level 3) within the time frame. |
| Derivation | Number of noc clinically signif hypoglycaemic (level 2) (<3.0 (54 mg/dL), corby BG meter) conocturnal sever hypoglycaemic (level 3) | ficant<br>episodes<br>mmol/L<br>nfirmed<br>or | From baseline<br>week 0 (V2) to<br>week 57 (V56) | umber of<br>isodes | Nocturnal hypoglycaemic episodes: episodes occurring between 00:01 and 05:59 both inclusive. |
| Derivation | Number of noc clinically signifully hypoglycaemic (level 2) (<3.0 (54 mg/dL), coby BG meter) | ficant<br>episodes<br>mmol/L | From baseline<br>week 0 (V2) to<br>week 57 (V56) | umber of isodes | Nocturnal hypoglycaemic episodes: episodes occurring between 00:01 and 05:59 both inclusive. |
| Derivation | Number of noc<br>severe hypogly<br>episodes (level | caemic | From baseline<br>week 0 (V2) to<br>week 57 (V56) | <br>imber of isodes | Nocturnal hypoglycaemic episodes: episodes occurring between 00:01 and 05:59 both inclusive. |
| Derivation | Achievement o<br>HbA <sub>1c</sub> <7.0% (y | | At week 52 (V54) | ount of<br>bject | Dichotomous outcome variable: $Yes$ : Participant achieved HbA <sub>1c</sub> <7.0% $No$ : Participant did not achieve HbA <sub>1c</sub> <7.0% Missing HbA <sub>1c</sub> data at 52 weeks will be imputed in the same way as in the primary analysis before deriving the dichotomous outcome. |
| Derivation | Achievement o<br>HbA <sub>1c</sub> <7.0% w | rithout | At week 52 (V54) | ount of bject | Dichotomous outcome variable: Yes: Participant achieved HbA <sub>1c</sub> |

<7.0% without severe or

hypoglycaemic episodes during

clinically significant

the prior 12 weeks

VV-CLIN-219732 1.0

severe (level 3) or

clinically significant

hypoglycaemic episodes

(level 2) (<3.0 mmol/L

(54 mg/dL), confirmed by BG meter) during the prior 12 weeks (yes/no)

| Statistical Analysis Plan Study ID: NN1535-4592 CONFIDEN | Date: Version: Status: Page: | 23 June 2022 N. 5.0 Final 21 of 27 | lovo Nordisk |
|---|---|---|---|
|---|---|---|---|

| | | | | No: Participant did not achieve HbA1c <7.0% or participant had a severe or clinically significant hypoglycaemic episode during the prior 12 weeks or participant had discontinued randomised treatment Missing HbA1c data at 52 weeks will be imputed in the same way as in the primary analysis before deriving the dichotomous outcome. |
|---|---|---|---|---|
| Derivation | Achievement of HbA <sub>1c</sub> <7.0% without severe hypoglycaemic episodes (level 3) during the prior 12 weeks (yes/no) | At week 52 (V54) | Count of subject | Dichotomous outcome variable: Yes: Participant achieved HbA <sub>1c</sub> <7.0% without severe hypoglycaemic episodes during the prior 12 weeks No: Participant did not achieve HbA <sub>1c</sub> <7.0% or participant had a severe hypoglycaemic episode during the prior 12 weeks or participant had discontinued randomised treatment Missing HbA <sub>1c</sub> data at 52 weeks will be imputed in the same way as in the primary analysis before deriving the dichotomous outcome. |
| Derivation | Achievement of HbA <sub>1c</sub> ≤6.5% (yes/no) | At week 52 (V54) | Count of subject | Dichotomous outcome variable: $Yes$ : Participant achieved $HbA_{1c} \le 6.5\%$ $No$ : Participant did not achieve $HbA_{1c} \le 6.5\%$ Missing $HbA_{1c}$ data at 52 weeks will be imputed in the same way as in the primary analysis before deriving the dichotomous outcome. |
| Derivation | Achievement of HbA <sub>1c</sub> ≤6.5% without severe (level 3) or clinically significant hypoglycaemic episodes (level 2) (<3.0 mmol/L (54 mg/dL), confirmed by BG meter) during the prior 12 weeks (yes/no) | At week 52 (V54) | Count of subject | Dichotomous outcome variable: Yes: Participant achieved HbA <sub>1c</sub> ≤6.5% without severe or clinically significant hypoglycaemic episodes during the prior 12 weeks No: Participant did not achieve HbA1c ≤6.5% or participant had a severe or clinically significant hypoglycaemic episode during the prior 12 weeks or participant had discontinued randomised treatment Missing HbA <sub>1c</sub> data at 52 weeks will be imputed in the same way as in the primary analysis before deriving the dichotomous outcome. |

| Statistical Analysis Plan Study ID: NN1535-4592 CONFI | Date: Version: Status: Page: | Novo Nordisk |
|---|---|---|
|---|---|---|

| Derivation | Achievement of HbA <sub>1c</sub> ≤6.5% without severe hypoglycaemic episodes (level 3) during the prior 12 weeks (yes/no) | At week 52 (V54) | Count of subject | Dichotomous outcome variable: Yes: Participant achieved HbA <sub>1c</sub> ≤6.5% without severe hypoglycaemic episodes during the prior 12 weeks No: Participant did not achieve HbA <sub>1c</sub> ≤6.5% or participant had a severe hypoglycaemic episode during the prior 12 weeks or participant had discontinued randomised treatment Missing HbA <sub>1c</sub> data at 52 weeks will be imputed in the same way as in the primary analysis before deriving the dichotomous outcome. |
|---|---|---|---|---|
| Derivation | Achievement of HbA <sub>1c</sub> <7.0% without body weight gain (yes/no) | At week 52 (V54) | Count of subject | Dichotomous outcome variable: $Yes$ : Participant achieved HbA <sub>1c</sub> <7.0% and change in body weight from baseline week 0 to week $52 \le 0$ kg $No$ : Participant did not achieve HbA <sub>1c</sub> <7.0% <b>or</b> participant had a change in body weight from baseline week 0 to week $52 > 0$ kg Missing HbA <sub>1c</sub> data at $52$ weeks will be imputed in the same way as in the primary analysis and missing body weight data will be imputed in the same way as in analysis of body weight before deriving the dichotomous outcome. |
| Derivation | Achievement of HbA <sub>1c</sub> <7.0% without body weight gain and severe (level 3) or clinically significant hypoglycaemic episodes (level 2) (<3.0 mmol/L (54 mg/dL), confirmed by BG meter) during the prior 12 weeks (yes/no) | At week 52 (V54) | Count of subject | Dichotomous outcome variable: $Yes$ : Participant achieved HbA <sub>1c</sub> <7.0% without severe or clinically significant hypoglycaemic episodes during the prior 12 weeks and change in body weight from baseline week 0 to week $52 \le 0$ kg $No$ : Participant did not achieve HbA1c <7.0% or participant had a severe or clinically significant hypoglycaemic episode during the prior 12 weeks or participant had discontinued randomised treatment or participant had a change in body weight from baseline week 0 to week $52 > 0$ kg |

Page:


| | | | | Missing HbA <sub>1c</sub> data at 52 weeks will be imputed in the same way as in the primary analysis and missing body weight data will be imputed in the same way as in analysis of body weight before deriving the dichotomous outcome. |
|---|---|---|---|---|
| Derivation | Achievement of HbA <sub>1e</sub> <7.0% without body weight gain and severe hypoglycaemic episodes (level 3) during the prior 12 weeks (yes/no) | At week 52 (V54) | Count of subject | Dichotomous outcome variable: $Yes$ : Participant achieved HbA <sub>1c</sub> <7.0% without severe hypoglycaemic episodes during the prior 12 weeks and change in body weight from baseline week 0 to week $52 \le 0$ kg $No$ : Participant did not achieve HbA <sub>1c</sub> <7.0% or participant had a severe hypoglycaemic episode during the prior 12 weeks or participant had discontinued randomised treatment or participant had a change in body weight from baseline week 0 to week $52 \ge 0$ kg Missing HbA <sub>1c</sub> data at $52$ weeks will be imputed in the same way as in the primary analysis and missing body weight data will be imputed in the same way as in analysis of body weight before deriving the dichotomous outcome. |
| Derivation | Achievement of HbA <sub>1c</sub> ≤6.5% without body weight gain (yes/no) | At week 52 (V54) | Count of subject | Dichotomous outcome variable: $Yes$ : Participant achieved HbA <sub>1c</sub> $\leq$ 6.5% and change in body weight from baseline week 0 to week $52 \leq 0$ kg $No$ : Participant did not achieve HbA <sub>1c</sub> $\leq$ 6.5% or participant had a change in body weight from baseline week 0 to week $52 > 0$ kg Missing HbA <sub>1c</sub> data at $52$ weeks will be imputed in the same way as in the primary analysis and missing body weight data will be imputed in the same way as in analysis of body weight before deriving the dichotomous outcome. |

| Statistical Analysis Plan | | Date: | 23 June 2022 Novo Nordisk |
|---|---|---|---|
| Study ID: NN1535-4592 | CONFIDENTIAL | Version: | 5.0 |
| | CONFIDENTIAL | Status: | Final |
| | | Page: | 24 of 27 |

| Derivation | Achievement of HbA <sub>1c</sub> ≤6.5% without body weight gain and severe (level 3) or clinically significant hypoglycaemic episodes (level 2) (<3.0 mmol/L (54 mg/dL), confirmed by BG meter) during the prior 12 weeks (yes/no) | At week 52 (V54) | Count of subject | Dichotomous outcome variable: Yes: Participant achieved HbA <sub>1c</sub> ≤6.5% without severe or clinically significant hypoglycaemic episodes during the prior 12 weeks and change in body weight from baseline week 0 to week 52 ≤ 0 kg No: Participant did not achieve HbA1c ≤6.5% or participant had a severe or clinically significant hypoglycaemic episode during the prior 12 weeks or participant had discontinued randomised treatment or participant had a change in body weight from |
|---|---|---|---|---|
| | | | | baseline week 0 to week 52 > 0 kg Missing HbA <sub>1c</sub> data at 52 weeks will be imputed in the same way as in the primary analysis and missing body weight data will be imputed in the same way as in analysis of body weight before deriving the dichotomous outcome. |
| Derivation | Achievement of HbA <sub>1c</sub> ≤6.5% without body weight gain and severe hypoglycaemic episodes (level 3) during the prior 12 weeks (yes/no) | At week 52 (V54) | Count of subject | Dichotomous outcome variable: <i>Yes</i> : Participant achieved HbA <sub>1c</sub> ≤6.5% without severe hypoglycaemic episodes during the prior 12 weeks and change in body weight from baseline week 0 to week 52 ≤ 0 kg <i>No</i> : Participant did not achieve HbA <sub>1c</sub> ≤6.5% or participant had a severe hypoglycaemic episode during the prior 12 weeks or participant had discontinued randomised treatment or participant had a change in body weight from baseline week 0 to week 52 > 0 kg Missing HbA <sub>1c</sub> data at 52 weeks will be imputed in the same way as in the primary analysis and missing body weight data will be imputed in the same way as in analysis of body weight before deriving the dichotomous outcome. |
| Derivation | Change in waist circumference | From baseline<br>week 0 (V2) to<br>week 52 (V54) | cm | The waist circumference value at baseline week 0 subtracted from the waist circumference value at week 52. |

 Date:
 25 Julie 2022

 Version:
 5.0

 Status:
 Final

 Page:

| Derivation | Change in systolic blood pressure | From baseline<br>week 0 (V2) to<br>week 52 (V54) | mmHg | The systolic blood pressure value at baseline week 0 subtracted from the systolic blood pressure value at week 52. |
|---|---|---|---|---|
| Derivation | Change in diastolic blood pressure | From baseline<br>week 0 (V2) to<br>week 52 (V54) | mmHg | The diastolic blood pressure value at baseline week 0 subtracted from the diastolic blood pressure value at week 52. |
| Derivation | Change in pulse | From baseline<br>week 0 (V2) to<br>week 52 (V54) | bpm | The pulse value at baseline week 0 subtracted from the pulse value at week 52. |
| Parameter | Cholesterol | At week 52 (V54) | mmol/L | |
| Parameter | High density lipoprotein (HDL) cholesterol | At week 52 (V54) | mmol/L | |
| Parameter | Low density lipoprotein (LDL) cholesterol | At week 52 (V54) | mmol/L | |
| Parameter | Very low density<br>lipoprotein (VLDL)<br>cholesterol | At week 52 (V54) | mmol/L | |
| Parameter | Triglycerides | At week 52 (V54) | mmol/L | |
| Parameter | Free fatty acids | At week 52 (V54) | mmol/L | |


Version: 5.0 Status: Final 26 of 27 Page:

#### 6.3 **Appendix 3: Attributable intercurrent events**

| Intercurrent event | Attributable | |
|---|---|---|
| Initiation of non-randomised insulin treats for more than 2 weeks | Yes | |
| Discontinuation of randomised treatment for any reason Adverse events possible or probable related to randomised treatment | | Yes |
| | Adverse events not possible or probable related to randomised treatment | No |
| | Hypoglycaemic episodes | Yes |
| | Included in the study in violation of the inclusion and/or exclusion criteria | Yes |
| | Simultaneous use of an approved or non-<br>approved investigational medicinal<br>product in another clinical study | Yes |
| | Lack of efficacy | Yes |
| Withdrawal of consent | | Yes |
| | Pregnancy or intention of becoming pregnant | No |
| | Other | No |

| Statistical Analysis Plan Study ID: NN1535-4592 CONFIDENTIAL | Date:<br>Version:<br>Status:<br>Page: | 23 June 2022 <b>Novo Nordisk</b> 5.0 Final 27 of 27 |
|---|---|---|
|---|---|---|

## 7 References

1. McEvoy BW. Missing data in clinical trials for weight management. J Biopharm Stat. 2016;26(1):30-6.

- 2. Little R, Rubin D. Statistical analysis with missing data. Sons. JW, editor. New York.: John Wiley & Sons. 1987.
- 3. Darken P, Nyberg J, Ballal S, Wright D. The attributable estimand: A new approach to account for intercurrent events. Pharm Stat. 2020;19(5):626-35.
- 4. Little RJA, Rubin DB. Statistical analysis with missing data. New York: Wiley. 1987. xiv, 278 p. p.